CLINICAL TRIAL: NCT01148524
Title: A Phase 2b/3, Multi-Center, Extension Study of V72P10 to Assess Antibody Persistence at Eighteen Months After the Completion of the Vaccination Course in Study V72P10.
Brief Title: Assessment of Antibody Persistence at Eighteen Months After the Completion of the Vaccination Course in Study V72P10
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P10E1
Record Dates: First submitted 2010-06-04; First posted 2010-06-22 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Meningococcal Disease; Meningococcal Meningitis
Keywords: Meningococcal disease; Vaccines; Adolescents
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

ARMS (9):
- rMenB06 (Other): Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 6 months) and placebo (at 1 and 2 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB0 (Other): Subjects who had received 1 dose of rMenB+OMV-NZ (at 0 month) and 3 doses of placebo (at 1, 2 and 6 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB016 (Other): Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 1 and 6 months) and 1 dose of placebo (at 2 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB01 (Other): Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 1 month) and placebo (at 2 and 6 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB026 (Other): Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 2 and 6 months) and 1 dose of placebo (at 1 month) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB02 (Other): Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 2 months) and placebo (at 1 and 6 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB012 (Other): Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 1 and 2 months) and 1 dose of placebo (at 6 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- rMenB6 (Other): Subjects who had received 1 dose of rMenB+OMV-NZ (at 6 months) and 3 doses of placebo (at 0, 1 and 2 months) in V72P10 study had a blood draw.
  Interventions: Biological: rMenB+OMV-NZ
- Naive (Other): An additional study group of naïve subjects that served as a baseline comparator for assessing antibody persistence in the vaccine groups and had blood draw for serological analyses at the time of enrollment.
  Interventions: Biological: No Vaccine

INTERVENTIONS:
Biological: No Vaccine
  Arms: Naive
Biological: rMenB+OMV-NZ — Subjects who had received either rMenB+OMV-NZ or placebo at study month 6 in V72P10 study had a blood sample drawn for serological analyses at 18 months later (-1/+3 months).
  Other Names: Serogroup B meningococcal recombinant vaccine
  Arms: rMenB0; rMenB01; rMenB012; rMenB016; rMenB02; rMenB026; rMenB06; rMenB6

SUMMARY:
This was a Phase 2b/3, multi-center, extension study of V72P10 to assess antibody persistence at 18 months after the vaccination course in study V72P10 (NCT00661713).

Subjects who participated in study V72P10, and who meet all other enrollment criteria for this extension study, and a group of naïve subjects (defined as subjects who had never received rMenB+OMV NZ or other experimental MenB vaccines) of similar age to the subjects who were eligible to participate in this extension study, performed one study visit in which a single blood sample was drawn for MenB serological analyses.

ELIGIBILITY:
Inclusion Criteria:

Informed consent was obtained from all the subjects before enrollment into the study after the nature of the study had been explained.

Inclusion criteria for naive subjects, newly enrolled:

1. Healthy adolescents, 13-19 years of age (the age window is defined as the first day the subject turns 13 years of age up to the day before the subject turns 20 years of age).
2. For Minor subjects:

   * subjects who had given their written assent and whose parent or legal guardians had given written informed consent at the time of enrollment, after the nature of the study had been explained.

   For Adult subjects:
   * subjects who had given their written informed consent at the time of enrollment, after the nature of the study had been explained.
3. Were available for the visit scheduled in the study.
4. Were in good health as determined by medical history, physical examination, clinical judgment of the investigator.

Inclusion criteria for subjects who participated in the V72P10 study (follow-on subjects):

1. For Minor subjects: (≤18 years of age)

   * subjects who had given their written assent and whose parent or legal guardians had given written informed consent at the time of enrollment, after the nature of the study had been explained.

   For Adult subjects: (older than 18 years of age)
   * subjects who had given their written informed consent at the time of enrollment, after the nature of the study had been explained.
2. Who had participated in the V72P10 study and had received their last vaccination 18 months (-30 + 90 days) before enrollment in V72P10E1.
3. Who had completed the vaccination course in study V72P10, according to the protocol.
4. Who had provided at least the blood sample one month after the last vaccination in V72P10 (blood sample at visit 6, month 7), according to the protocol.
5. Were available for the study visit scheduled in the study.
6. Were in good health as determined by medical history, physical examination, clinical judgment of the investigator.

Exclusion Criteria:

Exclusion criteria for naïve subjects newly enrolled:

1. For Minor subjects:

   * subjects who were unwilling or unable to give written informed assent to participate in the study, and whose parent(s)/legal guardian(s) were unwilling or unable to give written informed consent to participate in the study

   For Adult subjects:
   * subjects who were unwilling or unable to give written informed consent to participate in the study.
2. History of any meningococcal B vaccine administration.
3. Previous ascertained or suspected disease caused by N. meningitidis.
4. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis.
5. Antibiotic treatment within 6 days prior to enrollment.
6. Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, diabetes mellitus Type I, cardiac disease, hepatic disease, neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition).
7. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids within 30 days prior to enrollment (use of low or moderate doses of inhaled steroids is not an exclusion);
8. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 90 days prior to enrollment.
9. Participation in another clinical trial within 90 days prior to enrollment or planned for during study.
10. Family members and household members of study staff.
11. Any condition which, in the opinion of the investigator, could have interfered with the evaluation of the study objectives.

Exclusion criteria for subjects who participated in the V72P10 study (follow-on subjects):

Exclusion criteria were the same as for naïve subjects, with the exception of criterion 2.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 817 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (6):
- Chile (6):
  - Centro de Salud Lo Barnechea, Santiago
  - Centro para vacunas en desarrollo. Hospital de Niños Roberto del Río, Santiago
  - Escuela de Medicina de la Universidad de Valparaíso, Santiago
  - Hospital Luis Calvo Mackenna, Santiago
  - Liceo Jose Victorino Lastarria, Santiago
  - Universidad de Chile. Facultad de Medicina, Santiago

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at six study sites in Chile.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- rMenB06: Subjects who had received 2 doses each of Recombinant Meningococcal B Vaccine with Outer Membrane Vesicle from the New Zealand Strain (rMenB+OMV-NZ) (at 0 and 6 months) and placebo (at 1 and 2 months) in V72P10 study.
- rMenB0: Subjects who had received 1 dose of rMenB+OMV-NZ (at 0 month) and 3 doses of placebo (at 1, 2 and 6 months) in V72P10 study.
- rMenB016: Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 1 and 6 months) and 1 dose of placebo (at 2 months) in V72P10 study.
- rMenB01: Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 1 months) and placebo (at 2 and 6 months) in V72P10 study.
- rMenB026: Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 2 and 6 months) and 1 dose of placebo (at 1 month) in V72P10 study.
- rMenB02: Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 2 months) and placebo (at 1 and 6 months) in V72P10 study.
- rMenB012: Subjects who had received 3 doses of rMenB+OMV-NZ (at 0, 1 and 2 months) and placebo (at 6 months) in V72P10 study.
- rMenB6: Subjects who had received 1 dose of rMenB+OMV-NZ (at 6 months) and 3 doses of placebo (at 0, 1 and 2 months) in V72P10 study.
- Naive: Age-matched subjects who had never received rMenB+OMV-NZ or other experimental MenB vaccines
Period: Overall Study
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive
Started | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51 | 151
Completed | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51 | 151
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled subjects.
Groups:
- rMenB06: Subjects who had received 2 doses each of rMenB+OMV-NZ (at 0 and 6 months) and placebo (at 1 and 2 months) in V72P10 study.
- Total: Total of all reporting groups
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive | Total
Number analyzed (Participants) | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51 | 151 | 817
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.2 (1.9) | 16.0 (2.0) | 16.2 (2.1) | 16.1 (1.9) | 15.6 (1.9) | 15.9 (1.8) | 15.9 (1.9) | 16.0 (1.9) | 15.6 (1.7) | 15.9 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 53 | 33 | 57 | 38 | 61 | 96 | 33 | 61 | 462
  Male | 19 | 42 | 20 | 45 | 19 | 45 | 57 | 18 | 90 | 355

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA Titers ≥1:4 Against Meningococcal Strains, At 18 Months After Month-6 Vaccination in V72P10 Study, and in Naive Subjects.
Description: The immune response was measured as the percentage of subjects with hSBA titers ≥1:4 against meningococcal strains 44/76-SL, 5/99 and NZ98/254, at 18 months after month-6 vaccination of rMenB+OMV-NZ or placebo in V72P10 study, and in age-matched vaccine naive subjects enrolled in this study, evaluated by serum bactericidal assay using human complement (hSBA).
Time Frame: month 0 (bl=baseline), month 1 and 18 months after last vaccination in V72P10 study.
Population: Analysis was performed on the modified intention-to-treat (MITT) data set, i.e. all subjects who provided evaluable serum samples. Samples were collected at 18 months post last vaccination in the parent study. For the Naive group, blood samples were obtained for meningococcal serology at day 1 and served as a comparator.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive
Number analyzed (Participants) | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51 | 151
Percentage of subjects
  S.44/76-SL-bl (N=49,95,53,102,57,106,153,51,0) | 31 [18 to 45] | 40 [30 to 51] | 40 [26 to 54] | 32 [23 to 42] | 32 [20 to 45] | 41 [31 to 51] | 44 [36 to 52] | 47 [33 to 62] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.44/76-SL-1m (N=49,95,53,102,57,106,153,51,0) | 100 [93 to 100] | 93 [85 to 97] | 100 [93 to 100] | 100 [96 to 100] | 100 [94 to 100] | 100 [97 to 100] | 100 [98 to 100] | 94 [84 to 99] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.44/76-SL-18m | 84 [70 to 93] | 73 [63 to 81] | 92 [82 to 98] | 82 [74 to 89] | 86 [74 to 94] | 81 [72 to 88] | 83 [76 to 89] | 73 [58 to 84] | 50 [42 to 59]
  S.5/99-bl (N=49,95,53,102,57,106,153,51,0) | 22 [12 to 37] | 33 [23 to 43] | 28 [17 to 42] | 26 [18 to 36] | 21 [11 to 34] | 30 [22 to 40] | 34 [27 to 42] | 33 [21 to 48] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.5/99-1m (N=49,95,53,102,57,106,153,51,0) | 98 [89 to 100] | 96 [90 to 99] | 100 [93 to 100] | 100 [96 to 100] | 100 [94 to 100] | 100 [97 to 100] | 100 [98 to 100] | 88 [76 to 96] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.5/99-18m | 94 [83 to 99] | 65 [55 to 75] | 98 [90 to 100] | 93 [86 to 97] | 100 [94 to 100] | 95 [89 to 98] | 96 [92 to 99] | 73 [58 to 84] | 25 [18 to 33]
  S.NZ98/254-bl (N=49,95,53,102,57,106,153,51,0) | 29 [17 to 43] | 31 [21 to 41] | 32 [20 to 46] | 24 [16 to 33] | 21 [11 to 34] | 30 [22 to 40] | 30 [22 to 38] | 29 [17 to 44] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.NZ98/254-1m (N=49,95,53,102,57,106,153,51,0) | 100 [93 to 100] | 94 [87 to 98] | 100 [93 to 100] | 100 [96 to 100] | 98 [91 to 100] | 100 [97 to 100] | 99 [96 to 100] | 92 [81 to 98] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.NZ98/254-18m | 86 [73 to 94] | 62 [52 to 72] | 98 [90 to 100] | 75 [65 to 83] | 96 [88 to 100] | 75 [66 to 83] | 86 [79 to 91] | 61 [46 to 74] | 40 [32 to 48]

2. Primary Outcome: Geometric Mean hSBA Titers Directed Against Meningococcal Strains, At 18 Months After Month-6 Vaccination in V72P10 Study, and in Naive Subjects.
Description: The immune response was measured as the hSBA geometric mean titers (GMTs) directed against meningococcal strains 44/76-SL, 5/99 and NZ98/254, at 18 months after month-6 vaccination of rMenB+OMV-NZ or placebo in V72P10 study, and in age-matched vaccine naive subjects enrolled in this study.
Time Frame: month 0 (bl=baseline), month 1 and 18 months after last vaccination in V72P10 study.
Population: Analysis was performed on the MITT data set.Samples were collected at 18 months post last vaccination in the parent study. For the Naive group, blood samples were obtained for meningococcal serology at day 1 and served as a comparator.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive
Number analyzed (Participants) | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51 | 151
Geometric mean titers
  S.44/76-SL-bl (N=49,95,53,102,57,106,153,51,0) | 2.83 [1.85 to 4.31] | 3.75 [2.75 to 5.12] | 3.56 [2.37 to 5.34] | 2.74 [2.04 to 3.68] | 2.76 [1.86 to 4.1] | 3.24 [2.43 to 4.34] | 3.86 [3.02 to 4.93] | 4.33 [2.86 to 6.56] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.44/76-SL-1m (N=49,95,53,102,57,106,153,51,0) | 227 [161 to 320] | 47 [36 to 60] | 316 [227 to 439] | 189 [149 to 241] | 265 [192 to 365] | 227 [179 to 287] | 253 [208 to 309] | 62 [44 to 86] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.44/76-SL-18m | 27 [16 to 45] | 16 [11 to 23] | 50 [30 to 83] | 29 [20 to 42] | 44 [27 to 73] | 34 [24 to 49] | 42 [31 to 56] | 19 [12 to 32] | 4.52 [3.52 to 5.82]
  S.5/99-bl (N=49,95,53,102,57,106,153,51,0) | 2.31 [1.62 to 3.3] | 2.65 [2.04 to 3.44] | 2.55 [1.81 to 3.6] | 2.22 [1.73 to 2.85] | 1.72 [1.23 to 2.39] | 2.36 [1.84 to 3.01] | 2.63 [2.14 to 3.23] | 2.67 [1.88 to 3.79] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.5/99-1m (N=49,95,53,102,57,106,153,51,0) | 802 [574 to 1121] | 63 [49 to 81] | 1181 [856 to 1630] | 445 [352 to 562] | 1105 [808 to 1510] | 727 [577 to 916] | 605 [499 to 735] | 68 [49 to 94] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.5/99-18m | 65 [43 to 98] | 7.1 [5.24 to 9.6] | 121 [82 to 180] | 40 [30 to 54] | 100 [68 to 146] | 43 [33 to 58] | 73 [57 to 92] | 9.85 [6.57 to 15] | 2.13 [1.73 to 2.63]
  S.NZ98/254-bl (N=49,95,53,102,57,106,153,51,0) | 2.66 [1.8 to 3.92] | 2.65 [1.99 to 3.53] | 3.68 [2.53 to 5.35] | 2.15 [1.63 to 2.82] | 2.15 [1.5 to 3.1] | 2.63 [2.01 to 3.44] | 2.75 [2.19 to 3.44] | 2.68 [1.82 to 3.93] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.NZ98/254-1m (N=49,95,53,102,57,106,153,51,0) | 154 [107 to 221] | 33 [25 to 43] | 174 [123 to 248] | 78 [60 to 100] | 170 [121 to 238] | 115 [89 to 148] | 129 [105 to 160] | 43 [30 to 62] | NA [NA to NA] — Data were not collected since the Naive subjects were enrolled in this study as comparator.
  S.NZ98/254-18m | 27 [17 to 43] | 8.71 [6.12 to 12] | 42 [26 to 66] | 17 [12 to 24] | 41 [26 to 64] | 19 [14 to 27] | 23 [18 to 31] | 9.16 [5.71 to 15] | 3.23 [2.52 to 4.14]

3. Primary Outcome: Geometric Mean Ratio at 18 Months After Month-6 Vaccination, Over Baselines at Month 0 and at One Month After the Last rMenB+OMV-NZ Vaccination in the V72P10 Study.
Description: The immune response was measured as the geometric mean ratio (GMRs) of hSBA GMTs against meningococcal strains 44/76-SL, 5/99 and NZ98/254 as follow: GMTs at 1 month after last vaccination to baseline GMTs; GMTs at 18 months after last vaccination to baselines GMTs; and GMTs at 18 months after last vaccination to GMTs at 1 month after last vaccination.
Time Frame: month 0 (baseline), month 1 and 18 months after last vaccination in V72P10 study.
Population: Analysis was performed on the MITT data set. Naive group was not reported for this endpoint since GMR data for this group were not collected (subjects were enrolled in this study and no GMT values at 1m and 18 m after last vaccination in V72P10 are available).
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6
Number analyzed (Participants) | 49 | 95 | 53 | 102 | 57 | 106 | 153 | 51
Geometric mean ratio
  S.44/76-SL (1 m postvaccination to baseline) | 80 [53 to 122] | 12 [9.18 to 17] | 89 [60 to 133] | 69 [52 to 92] | 96 [65 to 141] | 70 [52 to 93] | 66 [52 to 83] | 14 [9.47 to 21]
  S.44/76-SL (18 m postvaccination to baseline) | 9.51 [5.93 to 15] | 4.26 [3.01 to 6.03] | 14 [8.95 to 22] | 11 [7.6 to 15] | 16 [10 to 25] | 11 [7.67 to 15] | 11 [8.2 to 14] | 4.46 [2.8 to 7.11]
  S.44/76-SL (18 m to 1 m postvaccination) | 0.12 [0.077 to 0.18] | 0.34 [0.25 to 0.47] | 0.16 [0.1 to 0.24] | 0.15 [0.11 to 0.21] | 0.17 [0.11 to 0.25] | 0.15 [0.11 to 0.21] | 0.16 [0.13 to 0.21] | 0.31 [0.2 to 0.48]
  S.5/99 (1 m postvaccination to baseline) | 347 [223 to 541] | 24 [17 to 33] | 462 [301 to 709] | 200 [147 to 273] | 644 [425 to 976] | 309 [227 to 419] | 230 [178 to 298] | 25 [16 to 39]
  S.5/99 (18 m postvaccination to baseline) | 28 [18 to 44] | 2.68 [1.94 to 3.7] | 47 [31 to 73] | 18 [13 to 25] | 58 [38 to 87] | 18 [14 to 25] | 28 [21 to 36] | 3.69 [2.39 to 5.7]
  S.5/99 (18 m to 1 m postvaccination) | 0.081 [0.055 to 0.12] | 0.11 [0.085 to 0.15] | 0.1 [0.071 to 0.15] | 0.091 [0.07 to 0.12] | 0.09 [0.063 to 0.13] | 0.06 [0.046 to 0.078] | 0.12 [0.096 to 0.15] | 0.15 [0.1 to 0.21]
  SNZ98/254 (1 m postvacc to baseline) | 58 [39 to 87] | 12 [9.22 to 17] | 47 [32 to 70] | 36 [27 to 48] | 79 [54 to 115] | 44 [33 to 58] | 47 [37 to 60] | 16 [11 to 24]
  S.NZ98/254 (18 m postvacc to baseline) | 10 [6.62 to 15] | 3.29 [2.41 to 4.5] | 11 [7.57 to 17] | 7.93 [5.89 to 11] | 19 [13 to 28] | 7.37 [5.5 to 9.88] | 8.42 [6.59 to 11] | 3.43 [2.25 to 5.2]
  S.NZ98/254 (18 m to 1 m postvaccination) | 0.17 [0.12 to 0.26] | 0.27 [0.2 to 0.35] | 0.24 [0.16 to 0.35] | 0.22 [0.17 to 0.29] | 0.24 [0.17 to 0.35] | 0.17 [0.13 to 0.22] | 0.18 [0.14 to 0.23] | 0.21 [0.14 to 0.31]

4. Primary Outcome: Geometric Mean Concentration Against Meningococcal 287-953 Antigen, At 18 Months After Month-6 Vaccination in V72P10 Study, and in Naive Subjects.
Description: The immune response was measured as the geometric mean concentrations (GMCs) directed against meningococcal 287-953 antigen, evaluated using enzyme-linked immunosorbent assay (ELISA), at 18 months after month-6 vaccination of rMenB+OMV-NZ or placebo in V72P10 study, and in age-matched vaccine naive subjects enrolled in this study.
Time Frame: 18 months after last vaccination V72P10 study.
Population: Analysis was performed on the MITT dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: UI/mL
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive
Number analyzed (Participants) | 35 | 34 | 35 | 35 | 35 | 35 | 35 | 34 | 35
UI/mL | 272 [186 to 397] | 55 [37 to 82] | 555 [376 to 818] | 217 [148 to 319] | 490 [333 to 721] | 150 [101 to 221] | 175 [119 to 256] | 59 [40 to 88] | 24 [20 to 27]

ADVERSE EVENTS:
Time Frame: 18 months after vaccination.
Description: There was no vaccine administered in the study. Only safety data related to the blood draw procedure were collected.
Arm/Group | rMenB06 | rMenB0 | rMenB016 | rMenB01 | rMenB026 | rMenB02 | rMenB012 | rMenB6 | Naive
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/95 | 0/53 | 0/102 | 0/57 | 0/106 | 0/153 | 0/51 | 0/151
Other Adverse Events (participants affected / at risk) | 0/49 | 0/95 | 0/53 | 0/102 | 0/57 | 0/106 | 0/153 | 0/51 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days